CLINICAL TRIAL: NCT04168229
Title: A Clinical Investigation of the Benefit of Directionality as a Function of Microphone Location: BTE Hearing Aids Versus ITE Hearing Aids
Brief Title: A Clinical Investigation of the Benefit: BTE Hearing Aids Versus ITE Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernafon AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BF003-1808
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: The study is a controlled, open-label, comparative trial using a cross-over design. The subjects first wore the BTE Hearing aids and then the ITE.
Who Masked: Outcomes Assessor
Masking Description: Masking is not possible as the differences in hardware between the devices is obvious. The subjects and Investigator will recognize which device is the new one and which is the comparator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITE Hearing Aid (Experimental): The subjects will wear the ITE devices in a field test for 10 +/-7 days. At the second and third visits they will perform speech testing in the lab in three randomized conditions (unaided, aided with ITE, and aided with BTE).
  Interventions: Device: Mermaid 9 ITE
- BTE Hearing Aid (Active Comparator): The subjects will wear the BTE devices in a field test for 10 +/-7 days. At the second and third visits they will perform speech testing in the lab in three randomized conditions (unaided, aided with ITE, and aided with BTE).
  Interventions: Device: Mermaid 9 BTE

INTERVENTIONS:
Device: Mermaid 9 ITE — A Hearing aid intended to amplify sounds and deliver them to the ear with a microphone and receiver housed in an in-the-ear hardware.
  Arms: ITE Hearing Aid
Device: Mermaid 9 BTE — A Hearing aid intended to amplify sounds and deliver them to the ear with a microphone and Receiver housed in a behind-the-ear hardware.
  Arms: BTE Hearing Aid

SUMMARY:
The current study will evaluate a new in-the-ear (ITE) hearing aid hardware. The goal is to evaluate the audiological performance, usability, feature function, and to identify unexpected or unwanted behaviour from the devices. The study plans to compare the behind-the-ear (BTE) hardware style with the ITE devices regarding the benefit received from different microphone locations.

DETAILED DESCRIPTION:
Hearing aids constantly undergo incremental improvements from already marketed devices. The new devices are expected to perform as well or better than the previous ITE devices.

The aim of the testing is to grant quality control prior to product launch according to Bernafon development requirements.

The current study will evaluate a new ITE hearing aid hardware. The firmware driving the hearing aid has already been sold on the market using the BTE hardware for almost one year and will now be launched using the ITE custom hardware. The goal is to evaluate the audiological performance, usability, feature function, and to identify unexpected or unwanted behaviour from the devices. The study plans to compare the two hardware styles regarding the benefit received from different microphone locations.

As human subjects are involved the validation falls under the definition of a clinical investigation. The validation will address the performance of the new chip using the ITE hardware, and ensure that there is no reduction in speech understanding between using the BTE and ITE hardware styles. Evaluating the overall performance of the Mermaid 9 ITE devices is important to validate that the end user is satisfied with the devices and that all user requirements are fulfilled. All features available in Mermaid 9 have been validated and are currently used on the market in Mermaid 9 BTE devices.

ELIGIBILITY:
Inclusion Criteria:

* All classifications of hearing loss (sensorineural, conductive, mixed)
* If the hearing loss is conductive or mixed it must be approved for amplification by a physician
* All shapes of hearing loss (flat, sloping, reverse slope, notch)
* Severity ranging from mild to severe
* German speaking
* Current hearing aid users
* Both genders
* Ages 18 and older
* Ability and willingness to sign the consent form

Exclusion Criteria:

* Contraindications for amplification
* Active ear disease
* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia, or other cognitive problems of the participant
* A reduced mobility making them unable to attend weekly study appointments
* Uncooperative so that it is not possible to record a valid pure tone audiogram
* A strongly reduced dexterity
* Central hearing disorders
* Bernafon employees
* Family members of Bernafon employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Speech Intelligibility Performance | Through study completion, an average of one month.
  Speech test scores will be measured with speech reception thresholds (SRTs) of speech in noise in three conditions: unaided, aided with the BTE device, and aided with the new ITE device. The test is the Oldenburg Sentence test (OLSA) and uses nonsense sentences. The score is measured by the the signal-to-noise ratio (SNR) at which 50% of words in a sentence list are correctly repeated. The speech is always presented at 65 decibels (dB) and the background noise varies to maintain the 50% correct. A lower SNR score indicates a better score. The maximum score will be 15 dB and the minimum will be -5 dB.
Word Recognition | Through study completion, an average of one month.
  Word recognition test scores will be measured with speech reception thresholds (SRTs) of speech in noise in three conditions: unaided, aided with the BTE device, and aided with the new ITE device. The test is called the Göttinger sentence test (GÖSA) and uses content relevant sentences that subjects repeat . The score is measured by the the signal-to-noise ratio (SNR) at which 50% of words in a sentence list are correctly repeated. The speech is always presented at 65 decibels (dB) and the background noise varies to maintain the 50% correct. A lower SNR score indicates a better score. The maximum score will be 15 dB and the minimum will be -5 dB.

SECONDARY OUTCOMES:
Subjective Performance of Aided Benefit | Through study completion, an average of one month.
  The subjective performance for the new device will be measured with the APHAB questionnaire (Abbreviated Hearing Aid Benefit Profile). The questionnaire is a list of 24 statement that the subjects must agree or disagree with using a scale of units from A to G (A being Always and G being Never). Each letter has a corresponding score used for the calculation: A receives 99, B receives 87, C receives 75, D receives 50, E receives 25, F receives 12, and G receives 1.
  An average for each subscale is calculated, and a global or overall score can be calculated by taking the mean of the three positive subscales (Ease of communication, Background noise, and Reverberation). For these three subscales a higher score indicates a better performance. The highest possible score is 99 and the lowest is 1. The fourth scale (Aversiveness) is a negative scale meaning that a higher score means a worse performance. The highest possible score is 99 and the lowest is 1.

OTHER OUTCOMES:
Adverse Events | Through study completion, an average of one month.
  The number of adverse events reported including adverse events (AEs) related to the device will be used to measure the outcome. Adverse Events will be collected in an interview with the subjects during the Appointment. The minimum number of adverse Events possible is 0 and the maximum is infinite. A lower number means a better Outcome.
Unexpected device behavior | Through study completion, an average of one month
  Subjects will a questionnaire to report unexpected behavior. A 5-point scale is used with 0 being the lowest answer possible (never occuring) and 5 being the highest answer possible (occuring often). A lower scale is a better score.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Simon, AuD, Principal Investigator — Bernafon AG
Locations (1):
- Bernafon AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT04168229/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04168229/SAP_001.pdf